CLINICAL TRIAL: NCT06134622
Title: Advancing Stroke Safety and Efficacy Through Early Tirofiban Administration After Intravenous Thrombolysis (ASSET-IT)
Acronym: ASSET-IT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Wei Hu, professor, The First Affiliated Hospital of University of Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASSET-IT
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Acute Ischemic Stroke
Keywords: tirofiban; intravenous thrombolysis
MeSH Terms: conditions — Ischemic Stroke | interventions — Tirofiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized, double-blind trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous thrombolysis plus tirofiban administration (Experimental): Patients will receive Intravenous thrombolysis and tirofiban administration
  Interventions: Drug: Intravenous thrombolysis plus tirofiban
- Intravenous thrombolysis plus placebo administration (Active Comparator): Patients will receive Intravenous thrombolysis and placebo (saline) administration
  Interventions: Drug: Intravenous thrombolysis plus placebo

INTERVENTIONS:
Drug: Intravenous thrombolysis plus tirofiban — Patients randomized to the Tirofiban group will receive continuous intravenous infusion of tirofiban for 24 hours: initial infusion of 0.4 μg/kg/min for 30 minutes followed by a continuous infusion of 0.1 μg/kg/min for up to 23.5 hours. The tirofiban placebo will be infused in a similar fashion.
  Arms: Intravenous thrombolysis plus tirofiban administration
Drug: Intravenous thrombolysis plus placebo — placebo (saline)
  Arms: Intravenous thrombolysis plus placebo administration

SUMMARY:
To assess the efficacy and safety of tirofiban administration after intravenous thrombolysis for patients with AIS.

DETAILED DESCRIPTION:
The standard treatment for acute ischemic stroke is intravenous thrombolysis to dissolve fibrin and restore blood flow. However, reocclusion of blood vessels and stroke progression remain challenges after this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Onset of ischemic stroke symptoms within ≤ 4.5 hours*, treated with intravenous rt-PA or TNK according to guidelines;
2. NIHSS score of 4-25 before intravenous thrombolysis;
3. Age ≥ 18 years;
4. Able to receive the designated study drug within 60 minutes after intravenous thrombolysis;
5. Informed consent signed by the patient or their legal representative. *Symptom onset is defined as the last known well time.

Exclusion Criteria:

1. Presence of contraindications to intravenous thrombolysis;
2. Pre-stroke mRS score > 1;
3. Patients planned to undergo mechanical thrombectomy or other endovascular treatments (e.g., intra-arterial thrombolysis);
4. Patients with a history of atrial fibrillation or emergency ECG indicating atrial fibrillation;
5. Pregnant or lactating women;
6. NCCT, CTA source imaging, or MRI-DWI showing ASPECTS or PC-ASPECTS < 6;
7. If NIHSS worsens by 2 or more points between start of thrombolysis and start of study drug, repeat brain imaging rules out new intracranial hemorrhage;
8. Severe leukoaraiosis;
9. Currently participating in other clinical trials;
10. Known genetic or acquired bleeding diathesis, or received warfarin and INR > 1.7; or treated with direct oral anticoagulant agents in the prior 48 hours;
11. Severe renal failure, defined as serum creatinine > 3.0 mg/dl (or 265.2 μmol/l) or glomerular filtration rate [GFR] < 30, or patients requiring hemodialysis or peritoneal dialysis;
12. Liver dysfunction (ALT > 2 times the upper limit of normal or AST > 2 times the upper limit of normal);
13. Known allergy to tirofiban or other IIb/IIIa inhibitors;
14. Life expectancy < 1 year;
15. Inability to complete 90-day follow-up (e.g., no fixed residence, overseas patients, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 832 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
a modified Rankin Score of 0-1 | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
mortality | 90 (± 14 days) after procedure
  (Number of subjects who died at 90-day follow-up/total number of subjects who participated in 90-day follow-up) x100%
symptomatic intracerebral hemorrhage (ICH) | within 36 hours after procedure
  SICH means any hemorrhage with neurological deterioration, as indicated by an NIHSS score that was higher by ≥4 points than the value at baseline or the lowest value in the first 36 hours or any hemorrhage leading to death.

SECONDARY OUTCOMES:
a modified Rankin Score of 0-3 | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Modified Rankin Score | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
NIHSS score | 24 hours after procedure
  The NIHSS is an ordinal hierarchical scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tao C, Liu T, Sun J, Zhu Y, Li R, Wang L, Zhang C, Song J, Jing X, Nguyen TN, Nogueira RG, Saver JL, Hu W. Advancing stroke safety and efficacy through early tirofiban administration after intravenous thrombolysis: The multicenter, randomized, placebo-controlled, double-blind ASSET IT trial protocol. Int J Stroke. 2025 Mar;20(3):373-377. doi: 10.1177/17474930241299666. Epub 2024 Nov 20. PMID 39501470
- [Derived] Tao C, Liu T, Cui T, Liu J, Li Z, Ren Y, Zhao X, Xie F, Li J, Wang H, Huang L, Li J, Wen J, Zeng J, Zhu J, Li Z, Li D, Hu X, Huang B, Wang J, Zhang C, Ye B, Hou Y, Gan Y, Sun H, Guan F, Shao Y, Liu Z, Ou Z, Fan S, Wang Y, Zhai H, Ni C, Wang H, Zhang C, Zhao Y, Wang G, Zhu Y, Li R, Sun J, Hu H, Cui J, Wang L, Zhang C, Song J, Jing X, Wang A, Wang J, Xu P, Qureshi AI, Nguyen TN, Nogueira RG, Saver JL, Hu W; ASSET-IT Investigators. Early Tirofiban Infusion after Intravenous Thrombolysis for Stroke. N Engl J Med. 2025 Sep 25;393(12):1191-1201. doi: 10.1056/NEJMoa2503678. Epub 2025 Jul 4. PMID 40616232